CLINICAL TRIAL: NCT01549847
Title: A Phase III, Randomized, Double Blind, Placebo Controlled Trial to Evaluate the Therapeutic Effect of the Association of L-carnitine and Piracetam as an Adjuvant Therapy in the Treatment of Weakness, Muscle Fatigue and Muscle Pain in the Postpoliomyelitis Syndrome
Brief Title: A Randomized, Double Blind, Placebo Controlled Trial L-carnitine and Piracetam in the Treatment of Weakness, Muscle Fatigue and Muscle Pain in the Postpoliomyelitis Syndrome
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was not approved by Health Surveillance Agency
Sponsor: Biolab Sanus Farmaceutica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAR-PIR.11.01
Record Dates: First submitted 2012-03-07; First posted 2012-03-09 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Postpoliomyelitis Syndrome
Keywords: Postpoliomyelitis Syndrome; Piracetam; L-Carnitine
MeSH Terms: conditions — Postpoliomyelitis Syndrome | interventions — Carnitine; Piracetam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- L-carnitine and piracetam (Experimental)
  Interventions: Drug: L-carnitine and piracetam
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: L-carnitine and piracetam — L-carnitine/piracetam (990mg/810mg) PO BID
  Arms: L-carnitine and piracetam
Drug: Placebo — Placebo PO BID
  Arms: Placebo

SUMMARY:
This protocol aims to assess of L-carnitine and piracetam to relieve weakness, muscle fatigue and muscle pain in patients with Postpoliomyelitis Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Postpoliomyelitis Syndrome diagnosis confirmed over a year;
* Electromyography test compatible with poliomyelitis;
* Preserved ability to swallow medication;
* Oral communication ability preserved;
* Preserved ability to perform pedaling test in at least one lower limb affected by Postpoliomyelitis Syndrome;
* Ability to understand information about the study and to document the decision about participating in the trial by signing the Informed Consent Form.

Exclusion Criteria:

* History of intolerance to L-carnitine or piracetam;
* Treatment with L-carnitine during the past 3 months;
* Treatment with piracetam or any other nootropics pyrrolidone derivatives, during the past three months;
* Anemia (hemoglobin reference range - men 13 to 17 g/dL and women 12 to 15 g/dL);
* High level of glycated hemoglobin (> 7.0%);
* Electrolyte imbalance (hypokalaemia - reference potassium concentration range: 3.5 to 5.6 mmol / L);
* Renal failure (creatinine reference range: 0.70 to 1.50 mg/dL);
* Urinary tract infection;
* Thyroid dysfunction (reference range: free T4: 0.54 to 0.67 mg/dL and TSH reference range: 0.5 to 5.5 μUI/mL) or usual treatment with thyroid hormone supplementation;
* Cardiomyopathy;
* Uncontrolled hypertension;
* Known or suspected autoimmune disease;
* Confirmed pregnancy, or plans to get pregnant during the trial;
* Depression or bipolar affective disorders with moderate to severe episodes within the last twelve months;
* Insulin-dependent diabetes mellitus;
* Treatment with anticoagulant drugs over two weeks (including non-steroidal anti-inflammatory drugs (NSAIDs), warfarin, phenprocoumon, heparin);
* Usual cocaine or alcohol use;
* Any other condition judged by the investigator as a possibility to interfere on the participant's decision to be part of the study or to accomplish investigation procedures.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
Changes in Muscle Weakness | 26 weeks
Changes in fatigue | 26 weeks

SECONDARY OUTCOMES:
Changes in muscle pain | 26 weeks
Changes in daytime sleepiness | 26 weeks
Changes in quality of life | 26 weeks
Changes in daily function | 26 weeks
Changes in depressive mood | 26 weeks
Changes in oxidative capacity in skeletal muscle | 26 weeks
Occurrence of adverse events | 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Acary Souza Bulle Oliveira, MD, PhD, Principal Investigator — Federal University of São Paulo
Locations (1):
- UNIFESP, São Paulo, São Paulo, Brazil